CLINICAL TRIAL: NCT06478862
Title: A Phase 2A Multicenter, Open Label Study of Promitil for the Treatment of Patients With Solid Tumors Associated With Deleterious Mutations Who Have Progressed After First Line Therapy
Brief Title: Promitil Treatment of Patients With Solid Tumors Associated With Deleterious Mutations Who Have Progressed After Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Lipomedix Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROM-2301
Record Dates: First submitted 2024-06-17; First posted 2024-06-27 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Cancer of Ovary; Pancreatic Ductal Adenocarcinoma
Keywords: Solid tumors; metastatic; inoperable; BRCA mutations
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: There will be 2 cohorts with up to 10 patients per cohort indication (ovarian/pancreatic). Eligible patients will be assigned in parallel to receive 6 cycles of Promitil treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pancreatic cancer (Experimental): Eligible subjects with pancreatic cancer will be intravenously (IV) administered 2.0 mg/kg Promitil on Day 1 of each 28-day cycle, for up to 6 cycles. Each cycle may be extended for up to 3 additional weeks (i.e., up to a total of 7 weeks from previous Day 1), if tolerability issues arise.
  Interventions: Drug: Promitil
- Ovarian cancer (Experimental): Eligible subjects with ovarian cancer will be intravenously (IV) administered 2.0 mg/kg Promitil on Day 1 of each 28-day cycle, for up to 6 cycles. Each cycle may be extended for up to 3 additional weeks (i.e., up to a total of 7 weeks from previous Day 1), if tolerability issues arise.
  Interventions: Drug: Promitil

INTERVENTIONS:
Drug: Promitil — The 10 patients recruited in each of the cohorts will receive intravenously (IV) administered 2.0 mg/kg Promitil on Day 1 of each 28-day cycle, for up to 6 cycles. Subjects who complete the 6-cycle Treatment Phase have the option to continue to receive Promitil until disease progression, death, unacceptable toxicity or withdrawal of consent.
  Other Names: Pegylated Liposomal Mitomycin-C Lipid-based Prodrug

SUMMARY:
This multicenter Phase 2a study was designed to evaluate the safety, tolerability, and efficacy of Promitil in patients with recurrent ovarian cancer and inoperable, locally advanced or metastatic pancreatic cancer, which bears deleterious germline or somatic mutations in BRCA1, BRCA2, or HRD (homologous recombination deficiency) -related genes.

Based on reported preclinical and clinical efficacy of Mitomycin C in BRCA-mutated tumors, and together with the demonstrated improved safety profile of Promitil in humans, it is expected that this liposomal formulation will have a favorable therapeutic index and significant clinical antitumor activity in patients with tumors bearing BRCA 1/2 and/or PALB2 mutations.

DETAILED DESCRIPTION:
The study will include a Screening, Treatment Phase and Long-Term Follow-up (LTFU) Phase. Upon signing the informed consent form, all subjects will undergo screening procedures to assess eligibility within 21 days prior to receiving study drug. Eligible subjects will be intravenously (IV) administered 2.0 mg/kg Promitil on Day 1 of each 28-day cycle, for up to 6 cycles. Subjects who complete the 6-cycle Treatment Phase have the option to continue to receive Promitil until disease progression, death, unacceptable toxicity or withdrawal of consent. During the 6-month Treatment Phase, safety assessments will be conducted at each study visit (Days 1, 2, 4,8 and 14 of Cycle 1, Day 1 of Cycle 2 and Cycles 4 and beyond and Days 1, 2 4,and 8 of Cycle 3). Safety will be assessed by measurement of weight, physical examinations, vital signs, ECG recordings, blood chemistry, hematologic and urinalysis parameters, and review of Adverse and Serious Adverse events (SAEs) and concomitant medications. Response will be assessed by CT/MRI/PET-CT scans and biomarker levels, with imaging conducted every 12 weeks (every 3 treatment cycles).For patients who stopped receiving Promitil for any reason other than disease progression, response will continue to be assessed every 12 weeks, until disease progression, death or withdrawal of consent, but no later than 1 year from first dose of Promitil. Once study treatment ends, all subjects will be followed up long-term, with survival status assessed every 3 months for up to 1 year or until death, the earlier of the two.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older on day of consent
2. Patient with either one of the following histologically or cytologically confirmed, deemed incurable malignancies:

   1. Recurrent ovarian cancer
   2. Inoperable, locally advanced or metastatic pancreatic ductal adenocarcinoma (PDAC)
3. Patient with PDAC measurable by RECIST 1.1. Previously irradiated lesions may be considered measurable if there has been demonstrated progression in these lesions. Ovarian cancer patients can have either measurable or non-measurable lesions (i.e., ovarian cancer patients with mostly ascites or pleural effusion are eligible)
4. Tumor with a known pathogenic or likely pathogenic germline or somatic mutation in BRCA1, BRCA2 or HRD-related genes as determined by a Clinical Laboratory Improvement Amendments (CLIA)-certified or equivalently accredited laboratory. Note: Patients with positive HRD score can be eligible regardless of any evidence for germline or somatic mutations
5. Patient received at least 1 line of chemotherapy for advanced pancreatic adenocarcinoma or ovarian cancer. Prior neoadjuvant and adjuvant chemotherapy are allowed, and platinum re-challenge is allowed for ovarian cancer patients for whom it is felt to be in their best interests, as determined by the Investigator. Prior PARP inhibitor, hormonal, biological, or immunological therapy are allowed. Palliative radiation therapy is allowed, provided it was/will be completed ≥2 weeks prior starting trial therapy
6. Capable of providing written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
7. ECOG performance status of 0 or 1
8. Adequate organ function as defined by:

   1. Absolute neutrophil count (ANC) ≥ 1500/µL
   2. Platelet count ≥ 100,000/µL
   3. Hemoglobin ≥ 9.5 g/dL
   4. Hematocrit ≥30%
   5. Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
   6. AST and ALT ≤ 3 x ULN OR ≤ 5 x ULN in the presence of liver metastases
   7. Albumin ≥ 3g/dL
   8. INR<1.5 unless on anticoagulants
9. Creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 45 mL/minute (as calculated by the Cockcroft-Gault formula)
10. Estimated life expectancy of at least 3 months
11. Patients (men and women) of reproductive potential willing and able to use an acceptable method of birth control as approved by the PI
12. With the exception of alopecia and neuropathy, resolution of all acute toxic effects of any prior chemotherapy, surgery or radiotherapy to NCI CTCAE (Version 5.0) Grade ≤ 1 or to the baseline laboratory values as defined in Inclusion Criteria Number 8 and 9.

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to, severe or ongoing active infection, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmias, or psychiatric illness/social situations that would limit compliance with study requirements
2. Any other severe concurrent disease which, in the judgment of the investigator, would make the subject unsuited for treatment
3. History of chronic active hepatitis, including carriage of hepatitis B virus (HBV) or hepatitis C virus (HCV), unless patient is adequately treated and shown to be serum virus-free
4. Evidence of active bleeding
5. Untreated brain metastases Note: Patients with brain metastases treated by surgery or radiation who are stable and symptom-free (≤ 4 mg dexamethasone/day) are eligible to participate in the study
6. Patient is pregnant or lactating
7. Prior intravenous treatment with MMC, either alone or in combination
8. Other anti-cancer treatment within 2 weeks before start of study drug
9. Other myelosuppressive treatment within 4 weeks before start of study drug
10. Treatment with other investigational drugs within 5 drug half-lives of day 1 of study drug
11. Patients with uncontrolled ascites that had more than one palliative abdominal tap up to 30 days prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-06-13 (Actual); Primary Completion 2026-01-02 (Actual); Study Completion 2026-01-02 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate at Month 6 | 24 weeks
  defined as the proportion of patients who are alive and without radiological or clinical progression, based on RECIST 1.1

SECONDARY OUTCOMES:
Incidence, severity, and duration of treatment-emergent adverse events (TEAEs) | 30 weeks
  TEAEs assessed by NCI Common Toxicity Criteria Adverse Events (CTCAE v5.0).
Objective response rate (ORR): | 24 weeks
  ORR: proportion of patients with partial or complete response (PR or CR, respectively), based on RECIST 1.1 criteria
Duration of response (DOR) | 24 weeks
  DOR: defined as the time from first evidence of confirmed objective response to the first occurrence of disease progression or death from any cause
Disease control rate (DCR) | 24 weeks
  DCR :defined as proportion of subjects alive and free of disease progression with either complete response (CR), partial response (PR) or stable disease (SD)
Overall survival (OS): | 52 weeks
  OS: time from first dose of Promitil to date of death from any cause
To assess the changes in tumor biomarker levels following treatment with Promitil | 24 weeks
  Changes from baseline in CA19-9, CA125, CA15.3 and/or CEA blood levels

OTHER OUTCOMES:
Plasma MLP (mitomycin lipidic pro-drug) level after Promitil infusion | 12 weeks
  Plasma MLP levels before and after each Promitil dose (1h, 4h, 24h, 4, 7days) as measured in cycles 1 and 3

CONTACTS AND LOCATIONS:
Overall Officials: Ora Rosengarten, MD, Principal Investigator — Shaare Zedek; Ofer Purim, MD, Principal Investigator — Shaare Zedek Medical Center; Ravit Geva, MD, Principal Investigator — Sourasky Medical Center; Amichai Meirovitz, MD, Principal Investigator — Soroka University Medical Center; Ruth Peretz, MD, Principal Investigator — Rambam Health Care Campus; Nirit Yarom, MD, Principal Investigator — Asaf Harofeh Medical Center; Tali Levy, MD, Principal Investigator — Wolfson Medical Center
Locations (6):
- Israel (6):
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Wolfson Medica Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - Shamir Medical Center (Asaf Harofeh), Ẕerifin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gabizon A, Shmeeda H, Tahover E, Kornev G, Patil Y, Amitay Y, Ohana P, Sapir E, Zalipsky S. Development of Promitil(R), a lipidic prodrug of mitomycin c in PEGylated liposomes: From bench to bedside. Adv Drug Deliv Rev. 2020;154-155:13-26. doi: 10.1016/j.addr.2020.07.027. Epub 2020 Aug 7. PMID 32777239
- [Background] Gabizon AA, Tahover E, Golan T, Geva R, Perets R, Amitay Y, Shmeeda H, Ohana P. Pharmacokinetics of mitomycin-c lipidic prodrug entrapped in liposomes and clinical correlations in metastatic colorectal cancer patients. Invest New Drugs. 2020 Oct;38(5):1411-1420. doi: 10.1007/s10637-020-00897-3. Epub 2020 Jan 18. PMID 31955309